CLINICAL TRIAL: NCT05253209
Title: A Phase III Double-Blind, Randomized, Placebo Controlled, Multi Center Clinical Study to Evaluate the Efficacy and Safety of Intravenous L-Citrulline for the Prevention of Clinical Sequelae of Acute Lung Injury Induced by Cardiopulmonary Bypass in Pediatric Patients Undergoing Surgery for Congenital Heart Defects
Brief Title: A Study Evaluating the Efficacy and Safety of IV L-Citrulline for the Prevention of Clinical Sequelae of Acute Lung Injury Induced by Cardiopulmonary Bypass in Pediatric Patients Undergoing Surgery for Congenital Heart Defects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim Analysis triggered futility
Sponsor: Asklepion Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIT-CPB-003-02
Record Dates: First submitted 2022-01-24; First posted 2022-02-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-08

CONDITIONS: Ventricular Septal Defect; Atrioventricular Septal Defect; Primum Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Atrioventricular Septal Defect; Partial atrioventricular canal | interventions — Citrulline; Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization via an IWRS. Study drug or placebo will be prepared and labeled with the appropriate subject identifiers only; no information that would reveal the contents of the dose to be administered (active versus placebo) will be included on the label. Study drug (citrulline or placebo) will be provided in either identical syringes or bags and mask labeled. The bags will be the same size, shape, and fluid clarity, and hence masked to both investigators and staff administering the drug. Only the pharmacist and the unblinded monitor responsible for performing drug accountability (a different monitor than the person performing routine data monitoring) will be aware of the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Patients will receive:
  1. an L-citrulline bolus of 150 mg/kg at the initiation of cardiopulmonary bypass
  2. the addition L-citrulline to maintain a steady state target concentration of approximately 100 μmol/L of L-citrulline during cardiopulmonary bypass
  3. an L-citrulline bolus of 10 mg/kg 30 minutes after decannulation from cardiopulmonary bypass, followed immediately by a 9 mg/kg/hour continuous L-citrulline infusion or placebo for up to 48 hours post-first dose. The infusion rate will be adjusted (up or down titration of drug infusion) to achieve a target steady state concentration of 100 μmol/L.
  Infusion will be discontinued once invasive arterial blood pressure monitoring is discontinued or at 48 hours, whichever occurs first.
  Interventions: Drug: L-citrulline
- Placebo (Placebo Comparator): Plasmalyte A administered to the same schedule as the active treatment arm.
  Interventions: Drug: Plasmalyte A

INTERVENTIONS:
Drug: L-citrulline — Intravenous L-citrulline given for up to 48 hours
  Arms: Active
Drug: Plasmalyte A — Intravenous Plasmalyte A given for up to 48 hours
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled, multicenter study to compare the efficacy and safety of L-citrulline versus placebo in patients undergoing surgery for congenital heart defects. Eligible patients undergoing repair of a large unrestrictive ventricular septal defect (VSD), a partial or complete atrioventricular septal defect (AVSD), or an ostium primum atrial septal defect (primum ASD) will be eligible for enrollment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, multicenter study that will compare the efficacy and safety of L- citrulline versus placebo in patients undergoing surgery for congenital heart defects. Eligible patients undergoing repair of a large unrestrictive ventricular septal defect (VSD), a partial or complete atrioventricular septal defect (AVSD), or an ostium primum atrial septal defect (primum ASD) will be eligible for enrollment.

Each enrolled patient will be randomized to receive either L citrulline or placebo throughout all administrations in the study. Patients will receive:

1. an L-citrulline bolus of 150 mg/kg or placebo at the initiation of cardiopulmonary bypass
2. the addition L-citrulline or placebo to maintain a steady state target concentration of approximately 100 μmol/L of L-Citrulline or placebo during cardiopulmonary bypass
3. an L-citrulline bolus of 10 mg/kg or placebo 30 minutes after decannulation from cardiopulmonary bypass, followed immediately by a 9 mg/kg/hour continuous L-citrulline infusion or placebo for up to 48 hours post-first dose. The infusion rate will be adjusted (up or down titration of drug infusion) to achieve a target steady state concentration of 100 µmol/L.

The study drug or placebo infusion will be discontinued once invasive arterial blood pressure monitoring is discontinued or at 48 hours, whichever occurs first. Patients will be followed until Day 28 or discharge from the hospital, whichever occurs first. For patients discharged prior to Day 28, a final assessment via telephone will be conducted at Day 28.

ELIGIBILITY:
Inclusion Criteria:

* Patients, parents, or legal guardian willing and able to sign informed consent
* Male and female subjects aged ≤18 years of age (females of child-bearing potential willing to practice an acceptable form of birth control)
* Patients undergoing cardiopulmonary bypass for repair of a large unrestrictive ventricular septal defect, an ostium primum/secundum atrial septal defect, or a partial or complete atrioventricular septal defect
* Pre-operative echocardiogram confirming cardiovascular anatomy and defect to be repaired

Exclusion Criteria:

* Evidence of pulmonary artery or vein abnormalities that will not be addressed surgically. Specific abnormalities excluded include:

  * significant pulmonary artery narrowing not amenable to surgical correction
  * previous pulmonary artery stent placement
  * significant left sided AV valve regurgitation not amenable to surgical correction
  * pulmonary venous return abnormalities not amenable to surgical correction
  * pulmonary vein stenosis not amenable to surgical correction
* Preoperative requirement for mechanical ventilation or IV inotrope support
* Presence of fixed or idiopathic pulmonary hypertension (i.e. Eisenmenger's Syndrome) prior to surgical repair
* Pre-operative use of medications to treat pulmonary hypertension
* Pregnancy; Sexually active females of child-bearing potential must be willing to practice an acceptable method of birth control for the duration of study participation (e.g. oral contraceptive, hormonal implant, intra-uterine device)
* Participation in another clinical trial within 30 days of Screening or while participating in the current study, including the 28 days of follow-up post study drug administration.
* Any condition which, in the opinion of the investigator, might interfere with the study objectives

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Post-operative need for mechanical ventilation | Time in hours from separation from CPB until discontinuation of all mechanical ventilation including non-invasive support or Day 28, whichever occurs first
  Mechanical ventilation is defined as invasive and non-invasive mechanical ventilation including bilevel positive airway pressure (BPAP), continuous positive airway pressure (CPAP)

SECONDARY OUTCOMES:
Intubation | From separation from bypass until discontinuation of intubation or Day 28, whichever occurs first
  Length of time on intubation
Early extubation | From end of surgery until 12 hours post-surgery
  Frequency of extubation <12 hours after surgery
Positive pressure ventilation | Time in hours from separation from CPB until discontinuation of all non-invasive mechanical ventilation or Day 28, whichever occurs first
  Length of time on non-invasive mechanical ventilation
Duration of hospitalization | From surgery until discharge from hospital or Day 28, whichever occurs first
  Number of post-operative days until discharge from hospital
Use of inotropes | Measured from first use until discharge or Day 28, whichever occurs first
  Duration of inotrope use (e.g., dopamine, dobutamine, milrinone, epinephrine, phenylephrine and/or norepinephrine).
Use of vasodilators | Measured from first use until discharge or Day 28, whichever occurs first
  Duration of vasodilator use (e.g., nitroprusside, nitroglycerin, and nicardipine)
Duration of chest tube placement | From the end of the surgery to the time the chest tube is removed or Day 28, whichever occurs first
  Total post-operative time chest tube is used
Volume of chest tube drainage | Duration of chest tube placement or Day 28, whichever occurs first
  Total amount of chest tube drainage (mL)
Hemodynamic improvement (heart rate) | 1, 2, 4, 12, 24, and 48 hours post-dose
  Changes in heart rate measurements.
Hemodynamic improvement (systemic arterial blood pressure) | 1, 2, 4, 12, 24, and 48 hours post-dose
  Changes in systemic arterial systolic and diastolic blood pressure measurements.
Hemodynamic improvement (oxygen saturation) | 1, 2, 4, 12, 24, and 48 hours post-dose
  Changes in oxygen saturation measurements.
Hemodynamic improvement (central venous pressure) | 1, 2, 4, 12, 24, and 48 hours post-dose
  Changes in oxygen saturation measurements.
Hemodynamic improvement (pulmonary arterial pressure) | 1, 2, 4, 12, 24, and 48 hours post-dose
  Changes in PAP measurements (when available).
Arterial blood gasses (PaO2) | Intra-operatively to Day 28
  Changes in PaO2 measurements
Arterial blood gasses (PaCO2) | Intra-operatively to Day 28
  Changes in PaCO2 measurements
Arterial blood gasses (HCO3) | Intra-operatively to Day 28
  Changes in HCO3 measurements
Arterial blood gasses (pH) | Intra-operatively to Day 28
  Changes in pH measurements
Plasma levels of L-citrulline to assess PK-PD (exposure-response) relationship | Pre-surgery, 6, 12, 24 and 48 hours after first dose
  Measurement of plasma levels of L-citrulline
Health Economics: mechanical ventilation | Total over duration of hospitalization or to Day 28 whichever occurs first
  Measured as cost per day and expressed as incremental cost per quality adjusted life year (QALY) gained
Health Economics: duration of hospitalisation | Total over duration of hospitalization or to Day 28 whichever occurs first
  Measured as total cost of hospitalisation expressed as incremental cost per quality adjusted life year (QALY) gained
Adverse events | Pre-operatively until Day 28
  Incidence of adverse events and serious adverse events
Incidence of refractory hypotension | From the end of surgery until 48 hours after first dose
  Number of subjects with any refractory hypotension. Defined as a drop of >20% in mean arterial pressure for >30 minutes.
Clinical laboratory values (Blood Hemoglobin and Total Bilirubin) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (Blood Haematocrit) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (Red Blood Cell Count) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (White Blood Cell Count) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (Blood Platelet Count) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (Blood Sodium, Potassium, Calcium, Magnesium, Chloride) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (Blood Urea Nitrogen and Creatinine) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (Blood Alkaline Phosphatase, Aspartate Aminotransferase, Alanine Aminotransferase) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (Blood Lactate Dehydrogenase) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.
Clinical laboratory values (Blood Activated Clotting Time) | Intra-operatively, Days 1, 2 and 28
  Absolute values and the absolute and percentage changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Mastropietro, MD, FCCM, Principal Investigator — Riley Hospital for Children at Indiana University Health; Gurdyal Kalsi, MD, MFPM, Study Director — Asklepion Pharmaceuticals, LLC
Locations (10):
- United States (10):
  - Children's of Alabama, Birmingham, Alabama
  - Children's Hospital of Colorado, Aurora, Colorado
  - Heart Center, Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Duke University Medical Center Surgical Office of Clinical Research (SOCR), Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital- The Heart Center, Columbus, Ohio
  - Seattle Children's Research Institute, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided